CLINICAL TRIAL: NCT03991234
Title: Improving the Academic Performance of First-Grade Students With Reading and Math Difficulty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Doug Fuchs, Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 180633
Record Dates: First submitted 2019-06-13; First posted 2019-06-19 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Reading Learning Disability; Math Learning Disability
MeSH Terms: conditions — Dyslexia; Dyscalculia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Coordinated Reading and Math Intervention (Experimental): Coordinated intervention provides 15 weeks (3 30-minute sessions per week) of explicit instruction addressing similar skills as those addressed in the reading intervention arm & similar skills as the math intervention arm.
  Interventions: Behavioral: Coordinated Intervention
- Reading Intervention (Active Comparator): Reading intervention provides 15 weeks (3 30-minute sessions per week) of explicit instruction designed to build skill on letter-sound associations, decoding, sight words, & contextualized reading.
  Interventions: Behavioral: Reading Intervention
- Math Intervention (Active Comparator): Math intervention provides 15 weeks (3 30-minute sessions per week) of explicit instruction on number knowledge, counting strategies, and arithmetic skill.
  Interventions: Behavioral: Math Intervention
- Business-as-usual Control (No Intervention): Participation in the school's typical reading and math classroom instruction and, if designated by the school, its supplemental program.

INTERVENTIONS:
Behavioral: Reading Intervention — Reading intervention provides 15 weeks (3 30-minute sessions per week) of explicit instruction to build skill on letter-sound associations, decoding, sight words, & contextualized reading.
  Arms: Reading Intervention
Behavioral: Math Intervention — Math intervention provides 15 weeks (3 30-minute sessions per week) of explicit instruction on number knowledge & counting strategies to build arithmetic skill.
  Arms: Math Intervention
Behavioral: Coordinated Intervention — Coordinated intervention provides 15 weeks (30-minute sessions per week) of explicit instruction addressing the similar skills as in the reading intervention arm & similar objectives as the math intervention arm.
  Arms: Coordinated Reading and Math Intervention

SUMMARY:
The main purpose of this clinical trials is to explore short-term effects of coordinated intervention versus the business-as-usual school program on the primary endpoints of post-intervention word-reading fluency and arithmetic fluency. The study population is students who begin 1st grade with delays in word reading and calculations. Students who meet entry criteria are randomly assigned to coordinated intervention across reading and math, reading intervention, math intervention, and a business-as-usual control group (schools' typical program). The 3 researcher-delivered interventions last 15 weeks (3 sessions per week; 30 minutes per session). Students in all 4 conditions are tested before researcher-delivered intervention begins and after it ends.

DETAILED DESCRIPTION:
First-grade students who meet study entry criteria are identified near the start of the school year using a 3-stage screening process. Students who enter the study complete the pretest battery.

Then, students are randomly assigned at the individual level to coordinated intervention, reading intervention, math intervention, or a business-as-usual control group (the schools' typical classroom instruction with supplemental intervention schools choose to provide). Research staff deliver intervention in the coordinated intervention condition, in the reading intervention condition, and in the math intervention condition 1:1 for 15 weeks (three 30-min sessions per week, scheduled in line with teacher input to avoid students missing important content). Adherence to the researcher-delivered interventions is monitored via audio recordings and live observations.

The content of each researcher-delivered intervention is aligned with the school district's 1st-grade foundational reading & math learning standards; relies on explicit instruction; and incorporates fluency-building activities word reading and/or arithmetic problems; incorporates procedures designed to build engagement and perseverance. Reading intervention is designed to build skill in letter-sound associations, decoding, sight words, and contextualized reading. Math intervention provides is designed to build number knowledge, counting strategies, and arithmetic skill. Coordinated intervention addresses the same instructional objectives as reading intervention & math intervention.

When researcher-delivered intervention ends, students in all four conditions complete the posttest assessment battery. Testers are blind to students' study conditions. Adherence to testing protocols is monitored via audio recordings. The primary endpoints are posttest word-reading fluency and arithmetic fluency.

ELIGIBILITY:
Inclusion Criteria:

* Attends a participating school in the Metropolitan-Nashville Public Schools
* Is a member of a first-grade classroom whose teacher has agreed to let his/her students participate
* Has the available school schedule to participate
* Has adequate English proficiency to be reliably assessed in English on study entry screening measures
* Scores at or below the 25th percentile on the study's screening math test
* Scores at or below the 25th percentile on the study's screening reading test
* Scores at or above the 7th percentile on at least one of the study's two measures of cognitive performance

Exclusion Criterion:

* Does not attend a participating school in the Metropolitan-Nashville Public Schools
* Is not a member of a first-grade classroom whose teacher has agreed to let his/her students participate
* Does not have the available school schedule to participate
* Does not have adequate English proficiency to be reliably assessed in English on study entry screening measures
* Scores above the 25th percentile on the study's screening math test
* Scores above the 25th percentile on the study's screening reading test
* Scores below the 7th percentile on both of the study's two measures of cognitive performance

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 383 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Word Reading Fluency-2 (Zumeta et al., 2012) | an average of 25 weeks
  Students have 1 min to read 60 words randomly sampled/presented in bands of 5 words from most frequent words; then from next-most frequent words; etc.). If students finish before 1 min, the score is prorated. Two alternate forms are administered.
Test of Word Reading Efficiency-Sight Word Efficiency | an average of 25 weeks
  The tester shows a word list ordered in increasing difficulty; children read as many words as they can in 45 seconds.
Arithmetic Combinations Fluency - Addition (Fuchs et al., 2013) | an average of 25 weeks
  Students have 1 minute to write answers to 25 addition items (sums 5-12).
Arithmetic Combinations Fluency - Subtraction (Fuchs et al., 2013) | an average of 25 weeks
  Students have 1 minute to write answers to 25 subtraction items (minuends 5-12).

SECONDARY OUTCOMES:
Wide Range Achievement Test-4-Reading (WRAT4; Wilkinson, & Robertson, 2006) | an average of 25 weeks
  Students read words ordered in difficulty (no time limit; testing ends after 10 consecutive errors).
WRAT-4-Arithmetic (Wilkinson, & Robertson, 2006) | an average of 25 weeks
  Children complete calculation problems of increasing difficulty (10 minutes).

OTHER OUTCOMES:
Comprehensive Test of Phonological Processing (CTOPP; Wagner et al., 2013)-Elision | an average of 25 weeks
  Students say words with a constituent part removed from the words.
CTOPP-Sound Matching | an average of 25 weeks
  Children see words and for each say which of 3 words (shown as pictures) start/end with the same sound.
SWAN Attentive Behavior Rating Scale (J. Swanson, 2004) | an average of 25 weeks
  Teachers rate 9 items from the DSM criteria for Attention Deficit Hyperactivity Disorder for inattention, each on a 7-point scale. The score is the sum of the 9 ratings.
The Grit Scale (Duckworth & Quinn, 2009)-grade 1 | an average of 25 weeks
  Students rate their own beliefs concerning perseverance in learning. The grade 1 adaptation simplifies language and situates questions entirely in terms of reading & math.
Rating Scale of Effort & Motivation (Malone & Fuchs, 2014) | an average of 25 weeks
  Teachers rate items assessing students' effort and motivation.
Working Memory Test Battery for Children - Nonword List Recall (WMTB-C; Pickering & Gathercole, 2001) | an average of 25 weeks
  Children repeat stimuli spoken by the tester in the same order. Trials correct is the score.
Test of First-Grade Reading Comprehension (Fuchs, Fuchs, Craddock, & Lehman, 2017). | an average of 25 weeks
  Children read short passages aloud and answer open-ended literal and inferential questions. Number correct is the score.
Test of First-Grade Math Word Problems (Fuchs, Seethaler, & Craddock, 2009) | an average of 25 weeks
  Children listen words problem read aloud to them, while they see the text, and find solutions.Number correct is the score.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Fuchs, Ph.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Research staff will make de-identified data sets electronically available to external users under a data-sharing agreement providing the user's commitment to use data for the research purposes described in the user's request; assurance that no research participant will be identified for any purpose; a commitment to securing the data; a commitment to not transferring data to other users & destroying the data after analyses are complete; & guarantees publications are credited to grant/agency and entered in PubMed. Once the user signs and returns the Agreement Form, a database with the variables of interest and codebook are provided, and staff provide relevant, de-identified data and segments of the code book with variable names/values, notes clarifying scoring/data-reduction methods not otherwise available, and a technical report describing the sample, study, and procedures.
Supporting Information: Study Protocol, SAP
Time Frame: The de-identified (stripped) primary outcome data set will become available no later than acceptance for publication of the main findings from the final data set and remain accessible for 3 years following the closeout of this grant. This time frame for data accessibility will be reviewed at the proposed project's completion and revised as needed.
  If all Investigators leave or become unavailable, the last remaining Investigator will assume responsibility for identifying a Vanderbilt faculty member to undertake these responsibilities.
Access Criteria: The user submits a request describing variables of interest, research aims, & quantitative methods and signs a user agreement form (see Plan Description).

DOCUMENTS (1):
  • Informed Consent Form (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT03991234/ICF_000.pdf